CLINICAL TRIAL: NCT04306094
Title: Predictive Prognostic Factors in Patients With Non-small Cell Lung Cancer Stage IV
Brief Title: Factors Determining the Prognosis in NSCLC Stage IV
Acronym: LUPROG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Ana Paula de Souza Borges, physician, MD, Instituto do Cancer do Estado de São Paulo
Other Study IDs: NP1105/17
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: NSCLC Stage IV
Keywords: prognostic factor; survival; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a cohort study with patients with advanced NSCLC. Patients will answer questionnaires about symptoms and quality of life and will be submitted to physical and blood tests, and computer tomography. The aim of this study is to estimate prognostic factors predicting survival to 3 months in patients with advanced NSCLC.

DETAILED DESCRIPTION:
Non-small-cell lung cancer (NSCLC) is currently the neoplasm leading in deaths worldwide and in Brazil. NSCLC has a high incidence, is usually diagnosed in advanced stages and has poor survival rates. The ability to refine the prognosis of a disease has implications at the time of diagnosis and decision about treatment. Clinical and laboratory factors are studied to evaluated the prognosis of diseases. Palliative Prognostic Score (PaP score), Karnofsky Performance Status Scale (KPS), Palliative Prognostic Index (PPI) are applied in patients with many types of solid tumors. The Charlson Score evaluates comorbidities and the attributed risk for presence it. Others predictors of prognostic are cachexia, quality of life, inflammatory factors, sarcopenia. There is a need to improve the ability to estimate the prognosis and to identify the factors responsible to low survival rates in patients with NSCLC diagnosed at advanced stage, also as a tool for a better treatment selection.

This is an observational and prospective study, including patients diagnosed with NSCLC and admitted in ICESP, staged as IV at admission, with no previous systemic treatment and classified as ECOG 2-4. Demographic data, presence of a caregiver, anthropometry, MRC dyspnea scale, KPS, Edmont Symptom Scale, Charlson's Comorbidity Score, PPI and PaP were evaluated in each patient. Evaluation of sarcopenia and cachexia with abdominal CT (Slice-O-Matic, v.5), arm circumference, handgrip strength test and quality of life using EORTC score QLQ C-30 and QLQ-CAX-24 were also evaluated. Significant prognostic factors will be selected by multivariate analysis in a training set estimated as 217 patients.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage IVa or IVb NSCLC patients histologically diagnosis.
* Eastern Cooperative Oncology Group Performance status 2 - 4
* Treatment-naive

Exclusion Criteria:

* Initiate treatment before initiate
* psychiatric illnesses, except depression
* pregnant or breastfeeding women
* two concomitant neoplasms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patient, treatment naive with Eastern Cooperative Oncology Group Performance status 2-4 (ECOG PS).
Sampling Method: Non-Probability Sample
Enrollment: 217 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 months
  to assess overall survival in patients with NSCLC

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Paula de Souza Borges, São Paulo, Brazil

REFERENCES:
- [Derived] Cunha MT, de Souza Borges AP, Carvalho Jardim V, Fujita A, de Castro G Jr. Predicting survival in metastatic non-small cell lung cancer patients with poor ECOG-PS: A single-arm prospective study. Cancer Med. 2023 Feb;12(4):5099-5109. doi: 10.1002/cam4.5254. Epub 2022 Sep 26. PMID 36161783